CLINICAL TRIAL: NCT05387135
Title: Transcutaneous Vagus Nerve Stimulation As a Pain Modulator in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Gehad Gamal Elsehrawy, Assistant Lecturer, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3905
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: Vagus nerve stimulation, knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham Transcutaneous Vagus Nerve Stimulation (Sham Comparator): For sham-t-VNS device was turned 180°, stimulating the outer earlobe which does not contain fibers of the ABVN. A similar protocol as for active stimulation was used.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- Transcutaneous Vagus Nerve Stimulation (Active Comparator): Afferents of the Auricular branch of vagus nerve (ABVN) were stimulated using a t-VNS device (TENS 7000TM) made by Roscoe Medical Inc., will be used. TENS 7000TM device was labeled as nerve stimulator and low-risk medical device (Instruction manual for TENS 7000). The electrode was placed in the left cymba concha with direct contact on the skin after cleaning with an alcohol swab. The stimulation for both groups will last for 30 minutes once a day for 3 days per week for 12 weeks. The amplitude of the output current was between 0.25-2.0 mA as tolerated and 250 µs width at 10 Hz.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — Afferents of the Auricular branch of vagus nerve (ABVN) were stimulated using a t-VNS device (TENS 7000TM made by Roscoe Medical Inc., will be used. TENS 7000TM device was labeled as nerve stimulator and low-risk medical device (Instruction manual for TENS 7000).

SUMMARY:
a single-blinded, randomized clinical trial, 68 patients divided into 2 groups: active and sham treatment. Afferents of the Auricular branch of vagus nerve are stimulated using a transcutaneous Vagus Nerve Stimulation device (TENS 7000TM). The electrode was placed in the left cymba concha with direct contact on the skin. The stimulation for both groups will last for 30 minutes once a day for 3 days per week for 12 weeks. The amplitude of the output current was between 0.25-2.0 mA as tolerated and 250 µs width at 25 Hz. All participants initially will be evaluated before and after intervention and 3 months after the end of the sessions.

DETAILED DESCRIPTION:
The included study population is 68.

* Group (1): (tVNS group): This group of study subjects will include 34 patients of knee osteoarthritis and will be subjected to tVNS.
* Group (2): (sham group): This group of study subjects will include 34 patients of knee osteoarthritis and will be subjected to sham treatment.

DESCRIPTION OF THE TECHNIQUE

Active treatment:

Afferents of the Auricular branch of vagus nerve were stimulated using a t-VNS device (TENS 7000TM made by Roscoe Medical Inc., will be used. TENS 7000TM device was labeled as nerve stimulator and low-risk medical device (Instruction manual for TENS 7000). The electrode was placed in the left cymba concha with direct contact on the skin after cleaning with an alcohol swab. The stimulation for both groups will last for 30 minutes once a day for 3 days per week for 12 weeks. The amplitude of the output current was between 0.25-2.0 mA as tolerated and 250 µs width at 10 Hz.

Sham procedure:

For sham-t-VNS device was turned 180°, stimulating the outer earlobe which does not contain fibers of the ABVN. A similar protocol as for active stimulation was used.

All participants initially will be evaluated before and after intervention and 3 months after the end of the sessions by the following:

OUTCOME MEASURES AND ASSESSMENT QUESTIONNAIRES

1. Visual analogue scale (VAS)
2. PainDETECT questionnaire
3. DN4 questionnaire
4. Radiological Imaging
5. Knee injury and Osteoarthritis Outcome Score
6. Hospital Anxiety Depression Scale
7. Physical Function Tests
8. Quantitative sensory testing
9. The Central Sensitization Inventory

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Adult over 18 years.
* People who were diagnosed.
* Reported pain on visual analogue scale (VAS)>4/10.
* Able to understand the informed consent.

Exclusion Criteria:

* Peptic ulcer
* Pace maker
* Asthma or severe chronic obstructive pulmonary disease
* Pregnancy.
* Cellulites, skin ulceration at area of therapy application.
* Inability to fulfill follow-up criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 3 months
  to describe pain on 0 to 10 scale

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 months
  for function and activity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Hefny, MD, Study Director — professor of physical medicine, rheumatology and rehabilitation; Nashwa K Elshaarawy, MD, Study Director — Assisstant professor of physical medicine, rheumatology and rehabilitation; Nermeen H Abdelmoneam, Ph.D, Study Director — lecturer of physical medicine, rheumatology and rehabilitation
Locations (1):
- Suez Canal University, Ismailia, Egypt

REFERENCES:
- [Derived] Elsehrawy GG, Ibrahim ME, A Moneim NH, Hefny MA, El Shaarawy NK. Transcutaneous vagus nerve stimulation as a pain modulator in knee osteoarthritis: a randomized controlled clinical trial. BMC Musculoskelet Disord. 2025 Jan 20;26(1):68. doi: 10.1186/s12891-025-08288-6. PMID 39828740